CLINICAL TRIAL: NCT02238756
Title: Phase I Safety and Tolerability Trial of Single and Repeat Doses of the RNA-based Adjuvant CV8102 Alone and in Combination With a Licensed Rabies Virus Vaccine in Healthy Adults
Brief Title: Safety and Tolerability of CV8102 Alone and in Combination With a Rabies Virus Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CV-8102-201; 2013-004514-18 (EudraCT Number)
Record Dates: First submitted 2014-09-04; First posted 2014-09-12 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Rabies
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CV8102 (Experimental)
  Interventions: Biological: CV8102
- Rabipur (Active Comparator)
  Interventions: Biological: Rabipur
- CV8102 + Rabipur (Experimental)
  Interventions: Biological: CV8102 + Rabipur

INTERVENTIONS:
Biological: CV8102 — Subjects will receive 2 intramuscular doses of CV8102 given 21 days apart
  Arms: CV8102
Biological: Rabipur — Subjects will receive 2 intramuscular doses of Rabipur given 21 days apart
  Arms: Rabipur
Biological: CV8102 + Rabipur — Subjects will receive 2 intramuscular doses of CV8102+Rabipur given 21 days apart
  Arms: CV8102 + Rabipur

SUMMARY:
The purpose of this clinical trial is to investigate the safety and tolerability of IM administered CV8102 and an IM administered combination of CV8102 and rabies vaccine in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Compliant with protocol procedures and available for clinical F/U until the protocol-defined end of the trial
2. Physical examination and laboratory results without clinically significant findings
3. Body Mass Index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2
4. Subjects must use reliable forms of contraception (barrier method with spermicidal agent or true abstinence) and must refrain from sperm donation during treatment and the 4-week F/U period after the last treatment.

Exclusion Criteria:

1. Use of any investigational or non-registered product (adjuvant, drug) other than CV8102 within 4 weeks preceding the administration of the CV8102, or planned use of any such agent during the trial period
2. Subject has received any licensed or non-licensed vaccines within 4 weeks prior to the administration of CV8102 alone or in combination with the licensed rabies vaccine or planned vaccinations during the trial period
3. Any treatment with immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of CV8102 alone or in combination with the licensed rabies vaccine. The use of inhaled and nasal steroids, as well as topical steroids outside the vaccination area, will be permitted
4. Any medically diagnosed or suspected immune deficient condition based on medical history and physical examination
5. History of autoimmune disease or suspected autoimmune disease based on medical history and physical examination that cannot be ruled out based on further examinations
6. Administration of immunoglobulins (Igs) and/or any blood products within the 3 months preceding the administration of CV8102 or licensed rabies vaccine
7. Acute disease at the time of enrolment. Acute disease is defined as the presence of any acute condition including but not limited to non-febrile or febrile common colds, urinary tract infections, inflammatory, allergic or traumatic conditions that may interfere with safety assessment of the investigational products
8. Presence or evidence of significant acute or chronic disease, in particular heart disease including coronary artery disease and chronic pulmonary diseases (e.g., chronic obstructive pulmonary disease [COPD]); uncontrolled medical or psychiatric illness (subjects with uncomplicated chronic diagnoses stable and treated for ≥ 3 months e.g., mild hypertension well-controlled with medication, may be enrolled - provided the condition and its therapy are known not to be associated with an immunocompromised state or an autoimmune disease)
9. Major congenital defects
10. Known allergy to any component (or closely related substance) of the licensed rabies vaccine product
11. Known type I allergy to beta-lactam antibiotics
12. Evidence of current alcohol or drug abuse
13. History of any neurological disorders or seizures
14. Known seropositivity for human immunodeficiency virus (HIV), hepatitis B virus (HBV) (except in subjects previously vaccinated against HBV) or hepatitis C virus (HCV)
15. Foreseeable non-compliance with protocol as judged by the Investigator
16. History of any life-threatening anaphylactic reactions
17. Subjects with impaired coagulation in whom an IM injection is contraindicated.

    Additional exclusion criteria for subjects participating in the (adjuvanted) rabies vaccination part:
18. Subject has previously received any investigational or licensed rabies vaccine
19. Intending to travel to regions/countries for which rabies vaccinations are recommended or where high risk of infection exists according to travel recommendations by the German Society of Tropical Medicine and International Health (DTG) during the trial and F/U period
20. Subject is taking chloroquine for malaria treatment or prophylaxis.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with serious and non serious adverse events | Up to 12 months

SECONDARY OUTCOMES:
Maximum tolerated dose (MTD) of CV8102 within the dose range of 25 µg to 250 µg. | Up to day 49
MTD of CV8102 in combination with rabies vaccine | Up to Day 49
Vaccination-elicited serum rabies VNTs among the dose groups | Up to day 35
Vaccination-elicited innate and adaptive immune responses | Up to Day 35
  Evaluation of corresponding serum and blood parameters (e.g. relevant cytokines, chemokines, immune effector molecules and lymphocyte phenotyping)

CONTACTS AND LOCATIONS:
Overall Officials: Ingo Meyer, MD, Principal Investigator — CRS Clinical Research Services Mönchengladbach GmbH
Locations (1):
- CRS Clinical Research Services Mönchengladbach GmbH, Mönchengladbach, Germany